CLINICAL TRIAL: NCT06556420
Title: Analisi Del Microbiota Nasofaringeo in Pazienti Con Infezioni Respiratorie
Brief Title: Analysis of Nasopharyngeal Microbiota in Patients With Respiratory Infections
Acronym: MINIPAR
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, De Maio Flavio, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6603
Record Dates: First submitted 2024-07-30; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Respiratory Infection
Keywords: microbiota faringeo, infezioni respiratorie
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- controls
- patients with S. pyogenes infection
- patients with other respiratory infections

SUMMARY:
Respiratory tract infections represent the most frequent infectious pathology in community environments and when of bacterial origin, imply a morbid state generally supported by a pathogenic bacterial species predominant on the commensal flora of the airways. Among the most frequent bacterial infections of the upper respiratory tract in pediatric age we find acute bacterial pharyngitis or pharyngotonsillitis caused by Streptococcus pyogenes (β-hemolytic group A), for which antimicrobial therapy is clearly indicated, and which manifests itself with an onset sudden fever. It should also be remembered that some forms of pharyngitis are caused by Chlamydia pneumoniae, Mycoplasma pneumoniae, Bordetella pertussis and Legionella, commonly responsible for lower respiratory tract infections but recently also associated with upper respiratory tract infections. In childhood, a viral or bacterial infection of the upper respiratory tract (in particular pharyngitis, laryngitis) can easily lead to an infection of the lower respiratory tract (pneumonia). In fact, the inflammatory process triggered by a previous infection, generally viral, determines an impairment of mucociliary clearance which facilitates the proliferation not only of pathogenic bacteria but also of the commensal bacterial flora, normally non-pathogenic. An altered local microbial flora can, therefore, contribute to the pathogenesis of new infections or itself be responsible for invasive infections. The microbiota of the upper airways may therefore be a further factor influencing the susceptibility, frequency and severity of acute respiratory diseases. The oropharyngeal microbiota is in fact made up of numerous bacterial species which, by colonizing this anatomical tract, interact with the mucosa of the pharynx and therefore with the immune system, contributing to the homeostasis of the upper respiratory tract and consequently also preserving the integrity of the lower respiratory tract. As observed for other anatomical sites, the composition of the oropharyngeal microbiota is conditioned by external events, among which we find the use of antibiotics or oral disinfectant drugs which can favor the development of pathogenic microorganisms. Characterizing the oropharyngeal microbiota in a state of acute and/or chronic respiratory infection could increase knowledge on the microbiological signature associated with such infections and ineffective antibiotic treatments. Greater knowledge of it, also with future corrective purposes, as has now been demonstrated for other body areas, could be of great help in reducing the risk of acute recurrent disease and/or chronic consequences.

DETAILED DESCRIPTION:
In recent years, the microbiota of the upper airways has emerged as a further factor influencing the susceptibility, frequency and severity of acute respiratory diseases. Greater knowledge of it, also with corrective purposes, as has now been demonstrated for other body areas, could be of great help in reducing the risk of acute recurrent disease and/or chronic consequences. The oropharyngeal microbiota is in fact made up of numerous bacterial species which, by colonizing this anatomical tract, interact with the mucosa of the pharynx and therefore with the immune system, contributing to the homeostasis of the upper respiratory tract and consequently also preserving the integrity of the lower respiratory tract. As observed for other anatomical sites, the composition of the oropharyngeal microbiota is conditioned by external events, among which we find the use of antibiotics or oral disinfectant drugs which can favor the development of pathogenic microorganisms. For this reason, characterizing the oropharyngeal microbiota in a state of acute and/or chronic respiratory infection could increase knowledge on the microbiological signature associated with such infections and ineffective antibiotic treatments to the point of becoming a factor used to prevent respiratory tract infections.

ELIGIBILITY:
Inclusion Criteria:

* age 0-20 years
* signs and/or symptoms of acute respiratory tract infection such as cold, pharyngitis, laryngitis, tracheitis, otitis, epiglottitis, laryngotracheitis, bronchitis and pneumonia.

Exclusion Criteria:

* antibiotic therapies in the last 30 days
* treatments with prebiotics or probiotics in the last 60 days (in particular containing Streptococcus salivarius)
* hormone therapies in the last 60 days
* local therapies in the last 60 days
* treatments with oral cavity disinfectants in the last 30 days
* presence of other pre-existing or ongoing respiratory pathologies
* current severe sepsis (sepsis criteria + organ dysfunction, peripheral hypoperfusion, hypotension)

Ages: 0 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who access the Pediatric Emergency Department with respiratory symptoms attributable to acute respiratory infection attributable to a bacterial and/or viral nature (diagnosed through nasopharyngeal swab as per normal clinical practice), who have given their informed consent to participate in this study. Subjects accessing the Pediatric Emergency Department who will perform a nasopharyngeal swab, as per normal clinical practice, with a negative result will also be included in the study as controls, considering the same exclusion criteria reported below. Informed consent will therefore be acquired upon entry to the Pediatric Emergency Department and in relation to the outcome of the nasopharyngeal swab the subjects will then be stratified into groups.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pharingeal microbiota | 24 months
  Characterization of the pharyngeal microbiome (alpha and beta diversity, relative and differential abundances) in patients with symptoms attributable to respiratory infections

SECONDARY OUTCOMES:
Differences in microbiota in patients with diverse respiratory infections | 24 months
  To compare the pharyngeal microbiome (alpha and beta diversity, relative and differential abundances) of patients with bacterial respiratory infections with that of patients suffering from respiratory infections of viral origin at the time of diagnosis (baseline).